CLINICAL TRIAL: NCT07298720
Title: Assessing Fluid-responsiveness Using Non-invasive Hybrid Diffuse Optics on Peripheral Muscle
Acronym: hDOS-CO
Status: Recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Institut de Ciències Fotòniques (ICFO) (Unknown)
Responsible Party: Principal Investigator, Jaume Mesquida, Senior Clinical Researcher, Corporacion Parc Tauli
Other Study IDs: CEIm 2024/3001; INN2024003 (Other Grant/Funding Number: Institut d'Investigació i Innovació Parc Taulí); CIR2023014 (Other Grant/Funding Number: Institut d'Investigació i Innovació Parc Taulí)
Record Dates: First submitted 2025-11-24; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness
Keywords: Fluid-responsiveness; Hemodynamic monitoring; Preload-responsiveness; Cardiac output
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical care patient: Critical care patients with their blood pressure invasively monitored through an arterial line
  Interventions: Other: Passive Leg Raising maneuver

INTERVENTIONS:
Other: Passive Leg Raising maneuver — The PLR will be performed using automatic bed adjustment: Starting from a semi-recumbent position, the lower limbs will be elevated to a 45° angle while the trunk will be moved from semi-recumbent to supine. After three minutes, subjects will be returned to the initial semi-recumbent position.

SUMMARY:
Proof-of-concept observational study including ICU patients undergoing a PLR maneuver. Local microvasculature will be assessed with the hDOS platform on the brachioradialis muscle, deriving the microvascular blood flow index (BFI) and tissue oxygen saturation (StO2). CO will be assessed via an invasive hemodynamic monitor based on pulse waveform analysis through the patient's arterial line. The correlation over time between CO and microvascular parameters, and the ability of microvascular variables for predicting a positive CO response (increase > 10%) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Invasive blood pressure monitoring through an arterial line

Exclusion Criteria:

* Patients with suspected pregnancy
* Intra-abdominal hypertension
* Elevated intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with their blood pressure invasively monitored through an arterial line
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
CO Response | During procedure
  The relative increase in % of the CO, from baseline during the PLR (at 60-120 seconds within the maneuver), will be calculated. Those subjects with a relative increase equal to or above 10% will be classified as CO-responders to the PLR. On the other hand, if the increase in CO during the PLR is below 10%, subjects will be classified as non-responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Taulí Hospital Universitari, Sabadell, Spain/ Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR